CLINICAL TRIAL: NCT02756325
Title: Quantitative MRI for Functional Imaging of the Testis: A New Methodology for Evaluation of the Infertile Male
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is no longer with the institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-01637
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Infertility
Keywords: Azoospermia, IVF, MRI
MeSH Terms: conditions — Infertility; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI (Experimental)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Imaging will be performed using a clinical whole-body MRI and a pelvic phased-array coil. No intravenous contrast will be administered. Sequences will include Diffusion weighted imaging (DWI), T2 mapping, arterial spin labeling, and spectroscopy. The acquisition is expected to take approximately one hour

SUMMARY:
Infertility-the inability to conceive despite one year of properly timed unprotected intercourse-is a common problem. Of all types of male factor infertility, non-obstructive azoospermia may be the most difficult for couples. Importantly, patients with non-obstructive azoospermia are asked to make difficult decisions in terms of reproductive choice; surgical attempts at identifying sperm (microdissection testicular sperm extraction) are often offered to these patients without a guarantee of being able to identify sperm. New methodologies in terms of evaluation of azoospermic males PRIOR to the couple embarking upon IVF are needed urgently. The other potential benefit of non-invasive determination of testis function and spermatogenesis would be the potential targeting of sperm extraction procedures. We hypothesize that quantitative MRI employing advanced functional metrics will be sensitive to functional and metabolic differences between subsets of azoospermic cases and will improve upon current characterization of patients with this condition. Moreover, it is believed that these techniques will provide complementary information, such that they may be combined in a synergistic fashion for targeted extraction methodologies.

DETAILED DESCRIPTION:
Of all types of male factor infertility, non-obstructive azoospermia may be the most difficult for couples. Azoospermia (both obstructive and non-obstructive) occurs in approximately 10-20% of all infertile males with non-obstructive azoospermia encompassing the majority of cases.

In this study, quantitative MRI will be investigated by employing advanced functional metrics for addressing these challenges. Specifically, diffusion-weighted imaging will be assessed, multi-echo T2 mapping, arterial-spin labeling, and spectroscopy. No intravenous contrast will be administered for purposes of this study. It is hypothesized that these techniques will be sensitive to functional and metabolic differences between subsets of azoospermic cases and will improve upon current characterization of patients with this condition. Moreover, it is believed that these techniques will provide complementary information, such that they may be combined in a synergistic fashion for targeted extraction methodologies.

The goal of this exploratory study is to investigate whether associations exist between quantitative MRI metrics and the previously noted features of testis architecture.

ELIGIBILITY:
Inclusion Criteria:

* Men with normospermia who are initiating testosterone replacement and are over 18 years of age will provide semen samples to NYU Fertility Center.

Exclusion Criteria:

* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study.
* All women are excluded as such patients do not have the relevant anatomy being considered in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Testis Function from Quantitative MRI | Six Months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Alukal, MD, Principal Investigator — NYU Langone Health